CLINICAL TRIAL: NCT05919472
Title: Effects of Oral Iron Supplementation Before vs. at Time of Vaccination on Immune Response in Iron Deficient Kenyan Women
Brief Title: Effects of Oral Iron Supplementation on Vaccine Response in Iron Deficient Kenyan Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nicole Stoffel (Other)
Collaborators: Swiss Federal Institute of Technology (Other); University of Oxford (Other)
Responsible Party: Sponsor-Investigator, Nicole Stoffel, Prof. Dr., ETH Zurich
Organization: ETH Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIVA_II
Record Dates: First submitted 2023-06-07; First posted 2023-06-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Iron Deficiency Anemia
Keywords: Iron deficiency; Anemia; Vaccine response; Women of reproductive age
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies; Anemia | interventions — COVID-19 Vaccines; Vi polysaccharide vaccine, typhoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-treatment group (Experimental): Participants assigned to this group will receive 200 mg oral iron on alternate days on study days 1-56.
  Interventions: Dietary Supplement: Oral iron supplementation (pre-treatment); Biological: COVID-19 vaccine; Biological: MenACWY vaccine; Biological: Typhim Vi vaccine
- Simultaneous treatment group (Experimental): Participants assigned to this group will receive placebo on alternate days on study days 1-28 and 200 mg oral iron on alternate days on study days 29-56.
  Interventions: Biological: COVID-19 vaccine; Biological: MenACWY vaccine; Dietary Supplement: Oral iron supplementation (simultaneous treatment); Biological: Typhim Vi vaccine
- Control group (Placebo Comparator): Participants assigned to this group will receive placebo on alternate days on study days 1-56.
  Interventions: Biological: COVID-19 vaccine; Biological: MenACWY vaccine; Biological: Typhim Vi vaccine

INTERVENTIONS:
Dietary Supplement: Oral iron supplementation (pre-treatment) — Iron supplements as 200 mg oral iron as FeSO4 given on alternate day on days 1-56
  Arms: Pre-treatment group
Biological: COVID-19 vaccine — Johnson & Johnson COVID- 19 (JJ COVID-19) vaccination given on day 28 to all participants
Biological: MenACWY vaccine — MenACWY vaccination given on day 28 to all participants
Dietary Supplement: Oral iron supplementation (simultaneous treatment) — Iron supplements as 200 mg oral iron as FeSO4 given on alternate day on days 28-56
  Arms: Simultaneous treatment group
Biological: Typhim Vi vaccine — Typhim Vi vaccination given on day 28 to all participants

SUMMARY:
Iron deficiency (ID) anemia (IDA) is a global public health problem, with the highest prevalence in Africa. Vaccines often underperform in low- and middle- income countries (LMIC), and undernutrition, including ID, likely plays a role. Recent studies have shown the importance of iron status in vaccine response. Intravenous iron given at time of vaccination improved response to yellow fever and COVID-19 vaccines in IDA Kenyan women. Whether oral iron treatment would have a similar beneficial effect on vaccine response is uncertain. Also, timing of oral iron treatment needs further investigation.

The co-primary objectives of this study are to assess 1) whether IDA in Kenyan women impairs vaccine response, and whether oral iron treatment improves their response; 2) the timing of oral iron treatment to improve vaccine response (prior to vaccination vs at time of vaccination).

We will conduct a double-blind randomized controlled trial in southern Kenya to assess the effects of iron supplementation on response to three single-shot vaccines: Johnson & Johnson COVID- 19 (JJ COVID-19), the quadrivalent meningococcal vaccine (MenACWY) and the typhoid Vi polysaccharide vaccine (Typhim Vi). Women with IDA will be recruited and randomly assigned to three study groups: group 1 (pre- treatment) will receive 100 mg oral iron as ferrous sulfate (FeSO4) daily on days 1-56; group 2 (simultaneous treatment) will receive matching placebo daily on days 1-28, and 200 mg oral iron as FeSO4 daily on days 29-56; and group 3 (control) will receive matching placebo daily on days 1-56. Women in all groups will receive the JJ COVID-19 vaccine, the MenACWY and the Typhim Vi vaccine on day 28. Cellular immune response and serology will be measured at 28 days after vaccination in all groups.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the trial
* Female aged 18-49 years
* Moderate anemia (Hb <110 g/L, but not severely anemic with Hb <80 g/L) • Iron deficient (ZnPP >40 mmol/mol haem)
* Anticipated residence in the study area for the study duration

Exclusion Criteria:

* Major chronic infectious disease (e.g., HIV infection);
* Major chronic non-infectious disease (e.g., Type 2 diabetes, cancer);
* Chronic medications;
* Use of iron-containing mineral and vitamin supplementation 2 weeks prior to study start;
* COVID-19 vaccine or confirmed COVID-19 infection within the past 2 years
* MenACWY vaccine in the past
* Typhoid vaccine in the past
* Pregnant (confirmed by rapid test during screening) or lactating.
* Malaria (confirmed by rapid test) à study start will be postponed

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
anti-spike (S1) immunoglobulin (IgG) and anti-receptor-binding domain (RBD) IgG concentrations against severe acute respiratory syndrome (SARS)-Coronavirus (COV)-2 [iU/ml] | Day 56
IgG concentration against meningococcal serogroups A, C, W, and Y (anti-MenACWY IgG) [iU/ml] | Day 56
IgG concentration against Typhoid [iU/ml] | Day 56

SECONDARY OUTCOMES:
Hemoglobin concentration (g/L) at baseline | Day 1
Hemoglobin concentration (g/L) at time of vaccination | Day 28
Hemoglobin concentration (g/L) at study end | Days 56
Zinc protoporphyrin concentration (µmol/mol heme) at baseline | Day 1
Zinc protoporphyrin concentration (µmol/mol heme) at time of vaccination | Day 28
Zinc protoporphyrin concentration (µmol/mol heme) at study end | Day 56
Plasma iron concentration (µg/mL) at baseline | Day 1
Plasma iron concentration (µg/mL) at time of vaccination | Day 28
Plasma iron concentration (µg/mL) at study end | Day 56
Total iron binding capacity at baseline | Day 1
Total iron binding capacity at time of vaccination | Day 28
Total iron binding capacity at study end | Day 56
Transferrin saturation (%) at baseline | Day 1
Transferrin saturation (%) at time of vaccination | Day 28
Transferrin saturation (%) at study end | Day 56
Plasma ferritin concentration (µg/L) at baseline | Day 1
Plasma ferritin concentration (µg/L) at time of vaccination | Day 28
Plasma ferritin concentration (µg/L) at study end | Day 56
Soluble transferrin receptor concentration (mg/L) at baseline | Day 1
Soluble transferrin receptor concentration (mg/L) at time of vaccination | Day 28
Soluble transferrin receptor concentration (mg/L) at study end | Day 56
C-reactive protein concentration (mg/L) at baseline | Day 1
C-reactive protein concentration (mg/L) at time of vaccination | Day 28
C-reactive protein concentration (mg/L) at study end | Day 56
Retinol binding protein concentration (µmol/L) at baseline | Day 1
Retinol binding protein concentration (µmol/L) at time of vaccination | Day 28
Retinol binding protein concentration (µmol/L) at study end | Day 56
Alpha-glycoprotein (AGP) concentration at baseline | Day 1
Alpha-glycoprotein concentration (g/L) at time of vaccination | Day 28
Alpha-glycoprotein concentration (g/L) at study end | Day 56
T-cell response assessed with an enzyme-linked immunosorbent assay (ELISA) detecting IFN-gamma produced by CD4+ and CD8+ T cell responses to SARS-CoV-2 peptides at study end | Day 56
COVID-19 specific T cell response measured in peripheral blood mononuclear cells by ELISpot assay quantifying specific cytokines' concentration. | Day 56
Typhim Vi specific B-cell response measured in peripheral blood mononuclear cells by ELISpot assay quantifying antibodies' and memory B cell concentration. | Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Simon Karanja, PhD, Principal Investigator — JKUAT
Locations (1):
- Msambweni County Referral Hospital, Msambweni, Kenya

IPD SHARING:
Plan to Share IPD: No